CLINICAL TRIAL: NCT00338299
Title: An Open-Label Pilot Study to Evaluate the Effects of Alternate Dosing of PROCRIT� (Epoetin Alfa) in the Treatment of Patients With Cancer and Chemotherapy Induced Anemia (60,000 Units Weekly for Four Weeks Followed by 60,000 Units Every Two Weeks)
Brief Title: Alternate Dosing of PROCRIT (Epoetin Alfa) in Patients With Cancer and Chemotherapy Induced Anemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Collaborators: Ortho Biotech Products, L.P. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR005098
Record Dates: First submitted 2006-06-16; First posted 2006-06-20 (Estimated); Last update posted 2011-05-23 (Estimated); Status verified 2010-04

CONDITIONS: Anemia; Chemotherapy
Keywords: Anemia; hemoglobin; chemotherapy; subcutaneous injection; Epoetin alfa
MeSH Terms: conditions — Anemia | interventions — Epoetin Alfa

INTERVENTIONS:
Drug: Epoetin alfa

SUMMARY:
The purpose of this study was to test the effectiveness and safety of PROCRIT (Epoetin alfa) at a higher starting dose (60,000 Units) once per week, followed by a less frequent dose (60,000 Units every two weeks) in patients with cancer and chemotherapy induced anemia.

DETAILED DESCRIPTION:
This was an open-label, non-randomized, multicenter pilot study where patients who were receiving chemotherapy for non-myeloid malignancy (cancer) with a baseline hemoglobin (Hb) <= 11 g/dL were enrolled. The primary objective of this pilot study was to estimate the hematologic responses for the dosing regimen of PROCRIT (Epoetin alfa), starting at a dose of 60,000 Units (U) administered subcutaneously (sc, under the skin) once per week (qw) for four weeks ("Phase A"), followed by a dose of 60,000 U every two weeks (q2w) ("Phase B") in patients with cancer and chemotherapy induced anemia. If, at any time during the study the Hb level rose to >13 g/dL, PROCRIT (Epoetin alfa) therapy was held until the Hb reached <=12 g/dL, then resumed at a reduced dose in both Phase A and Phase B. The dose was also reduced if a very rapid Hb response occurred (i.e. an increase of more than 1.3 g/dL in a 2-week period). The secondary objective of the study was to determine the incidence of anti-erythropoietin antibodies (anti-EPO Ab), at baseline and at end of study/early withdrawal in patients who had received a minimum of one dose of PROCRIT (Epoetin alfa). Rarely, anti-erythropoietin antibodies may form in patients who have some types of diseases (e.g., autoimmune diseases, rheumatoid arthritis, anemia of chronic disease), or in response to exposure to erythropoietin products such as Epoetin alfa necessitating discontinuation of the erythropoietin agent and medical treatment that may include blood transfusions.

Safety evaluations included clinical laboratory tests (hemoglobin and hematocrit), vital signs measurements (blood pressure), and incidence and severity of adverse events.

This study determined if higher initial weekly doses resulted in a higher initial response rate and/or a more brisk hemoglobin rise. Patients received PROCRIT (Epoetin alfa) 60,000 Units (U) once a week for 4 weeks. At Week 5 if hemoglobin increased by >= 1 g/dL above baseline, the PROCRIT dose was changed to 60,000 U every 2 weeks for <= 12 weeks. An additional PROCRIT dose was given if chemotherapy completed before Week 16.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of non-myeloid malignancy (no history of myelodysplasia allowed) with a baseline hemoglobin of <= 11 g/dL, planned to receive chemotherapy for a minimum of 12 weeks
* Life expectancy of >= 6 months with an Eastern Cooperative Oncology Group (ECOG) Performance Status 0 - 2
* Negative serum pregnancy test at Screening and adequate contraceptive during treatment and for three months after treatment
* Adequate hematologic function, adequate renal function and adequate hepatic function.

Exclusion Criteria:

* Planned radiation during the study
* Anemia due to factors other than cancer/chemotherapy (i.e., iron, B12 or folate deficiencies, hemolysis or gastrointestinal bleeding)
* Prior treatment with Epoetin alfa or any other erythropoietic agent (e.g., Darbepoetin alfa) within the previous three months
* Significant, uncontrolled disease/dysfunction of the pulmonary, cardiovascular, endocrine, neurologic, gastrointestinal, or genitourinary systems not attributable to underlying malignancy or chemotherapy, uncontrolled hypertension or history of uncontrolled cardiac arrhythmias, pulmonary embolism, thrombosis
* Transfusion of platelets or packed red blood cells within 28 days prior to the first dose of study medication
* Planned stem cell harvest of bone marrow or high dose chemotherapy with stem cell transplant during study duration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2003-08; Study Completion 2004-04 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with a >= 1 g/dL increase in Hb above baseline in Phase A independent of transfusion within 4 weeks

SECONDARY OUTCOMES:
Phase B: Maintain or increase the absolute Hb level achieved in Phase A (up to 0.9 g/dL higher) or maintain or increase the Hb level above that achieved in Phase A independent of transfusion within 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- See also: An Open-Label Pilot Study to Evaluate the Effects of Alternate Dosing of PROCRIT� (Epoetin Alfa) in the Treatment of Patients with Cancer and Chemotherapy Induced Anemia (60,000 Units Weekly for Four Weeks Followed by 60,000 Units Every Two Weeks) — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=633&filename=CR005098_CSR.pdf
- See also: |Reddy PK; Williams D; Wilhelm FE. An Open-Label Pilot to Evaluate a Flexible Dosing Regimen of Epoetin Alfa for the Treatment of Chemotherapy-Induced Anemia: 60,000 Units Weekly Followed by 60,000 Units Every 2 Weeks — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=633&filename=CR005098_SupportiveCancerTherapy.pdf